CLINICAL TRIAL: NCT05709717
Title: Regenerative Therapy With Autologous Stromal Vascular Fraction Derived Mesenchymal Stem Cells and Platelet-rich Plasma to Treat Complex Perianal Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: SVF-PRP
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Perianal Fistula; Perianal Crohn Disease; Anal Fissure; Rectovaginal Fistula; Perianal Fistula Due to Crohn's Disease
MeSH Terms: conditions — Fissure in Ano; Rectovaginal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Regenerative therapy with SVF-PRP to supplement perianal surgery — Regenerative therapy with autologous stromal vascular fraction derived mesenchymal stem cells and platelet-rich plasma to supplement perianal surgery
  Other Names: SVF-PRP

SUMMARY:
Consecutive patients with complex anal fistula were prospectively followed for 12 months. Routine MRI was performed before and at 4 and 12 months after surgery. Continence was assessed likewise using a validated questionnaire. Fistula were drained with setons prior surgery. SVF was harvested from subcutaneous abdominal fat and PRP from peripheral blood. Distal fistulectomy to the sphincter was performed and the wound left open, while the internal orifice was closed. SVF-PRP was injected around the fistula. Patients showered their excision wound until dry. Outcomes were reported as median & interquartile range (IQR)

ELIGIBILITY:
Inclusion Criteria:

Perianal fistula Perianal fissure Anovaginal fistula Rectovaginal fistula Perianal Crohn's disease

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with complex perianal disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Healing | 1 year
  Absence of fistula opening and discharge, well-being
MRI healing | 1year
  Absence of active fistula and abscess

SECONDARY OUTCOMES:
Fecal continence | 1 year
  Vaizey score
Quality of life (general and related to perianal diseases) | 1 year
  FIQoL
Costs | 1 year
  Direct cost to patient, institution, and payee

CONTACTS AND LOCATIONS:
Overall Officials: Michel Adamina, MD, PD, MSc, EMBA HSG, Principal Investigator — Chief of Colorectal Surgery
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data could be shared upon reasonable request and pending ethical clearance